CLINICAL TRIAL: NCT00004832
Title: Randomized Study of 3,4-Diaminopyridine for Lambert-Eaton Myasthenic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Duke University (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13441; DUMC-577; DUMC-FDR001068
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-07

CONDITIONS: Lambert-Eaton Myasthenic Syndrome
Keywords: Lambert-Eaton myasthenic syndrome; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Amifampridine

INTERVENTIONS:
Drug: 3,4-diaminopyridine

SUMMARY:
OBJECTIVES: I. Evaluate the safety and effectiveness of 3,4-diaminopyridine (DAP) in the treatment of patients with Lambert-Eaton myasthenic syndrome (LEMS).

II. Determine the side-effects and benefits associated with DAP.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are randomized to receive 3,4-diaminopyridine (DAP) or placebo orally 3 times daily for 5 days, after which treatment is discontinued and patients are observed for at least 24 hours. At the end of the blinded study, patients may then elect to take open label DAP orally 3 times daily for 6 months; those who do so are monitored for clinical effects and side effects for at least 6 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Lambert-Eaton myasthenic syndrome (LEMS) based on weakness that predominates in proximal limb muscles and electromyography (EMG) findings of small amplitude muscle responses to nerve stimulation, which decrease further during nerve stimulation at 5 Hz and which increase at least 2-fold after maximum voluntary contraction of the muscle for 10-20 seconds Quantified Myasthenia Gravis (QMG) clinical score at least 5 --Prior/Concurrent Therapy-- Chemotherapy: No concurrent chemotherapy Endocrine therapy: Patients receiving immunosuppressants must be on the same dose of medication for at least 3 months prior to study entry Radiotherapy: No concurrent radiotherapy Surgery: No concurrent surgery Other: Patients receiving cholinesterase inhibitors must discontinue the medication at study entry if possible, or else be on the same dose of medication for at least 1 month prior to study entry --Patient Characteristics-- Hematopoietic: No significant hematologic disease Hepatic: No significant hepatic disease Renal: No significant renal disease Cardiovascular: No cardiac arrhythmia or significant cardiac disease Neurologic: No seizure disorder Other: Not pregnant Negative pregnancy test required of fertile women Effective contraception required of fertile women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 1994-08; Study Completion 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Donald B. Sanders, Study Chair — Duke University